CLINICAL TRIAL: NCT05249478
Title: A Comparative Study Between Continuous Epidural Analgesia Versus Ultrasound Guided Continuous Femoral Nerve Block (CFNB) Versus Ultrasound Guided Continuous Adductor Canal Block (ACB) for Post-operative Pain Management After Total Knee Replacement (TKR).
Brief Title: Pain Management After Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, remon nadhy, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ain Shams Universirty
Record Dates: First submitted 2021-11-25; First posted 2022-02-21 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
Keywords: epidural , adductor canal block, femoral nerve block, total knee replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- epidural catheter inserted before spinal anesthesia. (Active Comparator): As for the epidural analgesia, it will be performed under complete aseptic precautions, by introducing a needle between the lumbar vertebrae at level of L3-L4 or L4-L5 and injecting anesthetic medication into the epidural space, via the epidural catheter inserted through the needle into the epidural space.
  A small amount of air (1 to 2 mL) may be injected into the epidural space, avoid injecting larger amounts of air as this may contribute to patchy anesthesia.
  Interventions: Procedure: bupivacaine and fentanyl
- ultrasound guided femoral nerve catheter inserted before spinal anesthesia. (Active Comparator): As for the femoral nerve block, it will be performed under complete aseptic precautions, using a transportable Sonosite M-Turbo ultrasound system with linear transducer placed on the femoral crease to obtain the images of the femoral nerve & artery.
  The needle used for the block will be an echogenic needle of 18 Gauge and 3.5 inches. Before proceeding, skin infiltration with local anesthesia will be done using a syringe containing 5ml of 1% lidocaine, Once the femoral nerve is visualized, the needle will be inserted in-plane in a lateral to medial orientation and advanced towards the nerve. Once the tip placed adjacent to the nerve, the catheter is introduced through it, then the needle is removed, the location of the catheter can be confirmed by visualization of the catheter and spread of local anesthetic (LA).
  Interventions: Procedure: bupivacaine and fentanyl
- ultrasound guided adductor canal block inserted before spinal anesthesia. (Active Comparator): As for the adductor canal block,using a transportable Sonosite M-Turbo ultrasound system with linear transducer placed perpendicular to the thigh at the midpoint between the anterior superior iliac spine and the base of the patella,The needle used for the block will be an echogenic needle of 18 Gauge and 3.5 inches. Before proceeding, skin infiltration with local anesthesia will be done using a syringe containing 5ml of 1% lidocaine, the saphenous nerve is identified as it lies adjacent proximally lateral then distally superior to the femoral artery. Saphenous nerve is followed distally as it becomes more superficial, traveling with an arterial branch just deep to the sartorius muscle. Using an in-plane approach, after negative aspiration, the tip of the needle is placed deep to the sartorius muscle, at the lateral border of the artery, Once the needle is in position, the catheter is introduced through it, then the needle is removed.
  Interventions: Procedure: bupivacaine and fentanyl

INTERVENTIONS:
Procedure: bupivacaine and fentanyl — bupivacaine and fentanyl will be infused through the catheter

SUMMARY:
Aim of this study is to compare post-operative analgesic efficacy of continuous epidural analgesia versus ultrasound guided continuous femoral nerve block and adductor nerve block after unilateral total knee replacement using 0.125% bupivacaine.

DETAILED DESCRIPTION:
All patients will be assessed preoperatively, and will be instructed to fast for 8 hrs. On arrival to the operation theatre, Intravenous access will be established, and Ringer's solution will be infused as a co-load fluid bolus. Monitors for non-invasive blood pressure, heart rate, electrocardiogram (ECG), and pulse oximetry (SpO2) will be used to monitor the perioperative vital parameters of patients.

Before the spinal anesthesia, the epidural catheter will be inserted, while the femoral and adductor canal catheters will be inserted under ultrasound guidance before spinal anesthesia according to patient group allocation by single operator.

Group A: As for the epidural analgesia, it will be performed under complete aseptic precautions, by introducing a needle between the lumbar vertebrae at level of L3-L4 or L4-L5 and injecting anesthetic medication into the epidural space, via the epidural catheter inserted through the needle into the epidural space.

The epidural needle (typically 18-gauge and 8.89 cm (3.5 inches) in length) is inserted in the midline of the patient's back, defined by the spinous processes at the chosen spinal level. A skin wheal is raised with 1% lidocaine using a 25-gauge needle in the midline of the spine, in the lower third to half of the interspace. The subcutaneous tissue is infiltrated with lidocaine and is continued through supraspinous ligament down to the interspinous ligament.

The epidural needle is inserted with stylet at a straight or slight cephalad angle or at steeper cephalad angle. The needle bevel is oriented cephalad while the patient is in a sitting position. The needle is advanced through the supraspinous ligament and into the interspinous ligament. A firmness in the tissue suggests that the tip of the needle is in the supraspinous or interspinous ligament. Lack of firmness may indicate a paraspinous position of the needle tip, and the needle should be adjusted.

Once the needle tip is anchored in the interspinous ligament, the stylet is removed and a loss of resistance (LOR) syringe containing air is attached. Intermittent or continuous gentle pressure is applied to the plunger with the dominant thumb, while advancing the needle slowly with the nondominant hand. The ligamentum flavum is a tougher structure than the interspinous ligament and is identified by increased resistance to injection as the needle is advanced. Once LOR occurs, needle advancement is stopped to avoid an unintentional dural puncture.

The tip of the epidural needle is now located in the epidural space. A small amount of air (1 to 2 mL) may be injected into the epidural space, avoid injecting larger amounts of air as this may contribute to patchy anesthesia.

Group B: As for the femoral nerve block, it will be performed under complete aseptic precautions, using a transportable Sonosite M-Turbo ultrasound system with linear transducer placed on the femoral crease to obtain the images of the femoral nerve & artery (femoral nerve lateral or posterolateral to femoral artery at the level of the femoral triangle).

The needle used for the block will be an echogenic needle of 18 Gauge and 3.5 inches. Before proceeding, skin infiltration with local anesthesia will be done using a syringe containing 5ml of 1% lidocaine, Once the femoral nerve is visualized, the needle will be inserted in-plane in a lateral to medial orientation and advanced towards the nerve. Once the tip placed adjacent to the nerve, the catheter is introduced through it, then the needle is removed, the location of the catheter can be confirmed by visualization of the catheter and spread of local anesthetic (LA). Then 5 mL of lidocaine 1% will be injected through the needle under ultrasound guidance to confirm placement and inject the rest of the bolus through the catheter while visualizing spread of LA after removal of the needle. The catheter is secured to the skin with a sterile dressing after applying a sterile surgical glue.

Group C: As for the adductor canal block, it will be performed under complete aseptic precautions, using a transportable Sonosite M-Turbo ultrasound system with linear transducer placed perpendicular to the thigh at the midpoint between the anterior superior iliac spine and the base of the patella, the adductor canal is roofed by sartorius muscle and bounded medially by adductor longus muscle and laterally by vastus medialis muscle.

The needle used for the block will be an echogenic needle of 18 Gauge and 3.5 inches. Before proceeding, skin infiltration with local anesthesia will be done using a syringe containing 5ml of 1% lidocaine, the saphenous nerve is identified as it lies adjacent proximally lateral then distally superior to the femoral artery. Saphenous nerve is followed distally as it becomes more superficial, traveling with an arterial branch just deep to the sartorius muscle. Using an in-plane approach, after negative aspiration, the tip of the needle is placed deep to the sartorius muscle, at the lateral border of the artery, Once the needle is in position, the catheter is introduced through it, then the needle is removed.

5 ml of LA will be injected through the needle under ultrasound guidance to confirm placement and inject the rest of the bolus through the catheter while visualizing spread of LA. The catheter is secured to the skin with a sterile dressing after applying a sterile surgical glue.

In the three groups, Rescue doses of intravenous fentanyl will be given intravenously (IV) to the patient if there is still pain during positioning, increments of 50 microgram fentanyl (0.5 microgram/kg) and sedation score will be assessed and recorded.

Spinal anesthesia will be administered in the sitting position under complete aseptic conditions using a 25-gauge Quincke needle through L3-L4 or L4-L5 intervertebral space with 2 to 3.5 ml of 0.5% heavy bupivacaine and 25 microgram fentanyl with injection rate of 0.2 mL/second.

After confirmation of the start of sensory block, the level of the sensory block will be documented, and surgery will be allowed to start.

During operation, if any patient felt discomfort from the position or from the surgery, increments of fentanyl will be given IV and total intraoperative fentanyl will be recorded, and the surgery time will also be documented.

* Patients will be observed for any complications either related to the procedure e.g.: hematomas or related to drugs injected e.g.: hypotension, bradycardia, fall in peripheral oxygen saturation, nausea, vomiting or any other adverse effect and will be managed along with proper systematic assessment to exclude serious causes for any vital sign derangement .
* In case of hypotension (drop of blood pressure ˃20% of baseline reading), 3 mg increments of a 30 mg of ephedrine diluted with 10 ml normal saline 0.9% will be given intravenously by titration according to the blood pressure, along with 250 to 500 mL Ringer acetate as a fluid bolus if not contraindicated.
* In case of bradycardia, when it is associated with hypotension or any signs of impaired perfusion, 0.01 mg/kg of atropine will be given IV and repeated if needed.
* In case of fall in peripheral SpO2, supplemental oxygen will be given to keep SpO2 above 94%.
* In case of postoperative nausea and vomiting (PONV), 4 mg of ondansetron diluted with 10 ml normal saline 0.9% will be given intravenously slowly over 10 minutes.
* Postoperatively, continuous infusion of 0.125% bupivacaine with fentanyl 2µg/ml will be started through PCA at a fixed rate of 5 ml/hr. in the three groups
* Patients will be observed, and data recording will be done at 0,1,6,12,24,36 and 48 hours for postoperative pain scores, hemodynamic changes (blood pressure, heart rate and respiratory rate) and side effects such as pruritis, urine retention, nausea, vomiting and excessive motor block that prevents safe assisted or unassisted early postoperative mobilization. And the requirement of analgesic doses for the first 24 hours after the surgery will be noted.
* Postoperative pain and opioid consumption will be assessed after regaining of sensation in the contralateral limb by using visual analog scale (VAS) and VAS more than 3 will be managed by top up dose of 5ml.

ELIGIBILITY:
Inclusion Criteria:

.American Society of Anesthesiologists physical status (ASA) is I to III. .Both genders. .More than 40 years old.

Exclusion Criteria:

.Major spine deformities. .Bleeding disorders and coagulopathy. .Infection at the injection site. .Allergy to local anesthetics. .Pre-existing myopathy or neuropathy. .Significant cognitive dysfunction. .Patient refusal to participate.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
pain score | 48 hours
  Visual analogue score from 0 to 10

SECONDARY OUTCOMES:
hemodynamic changes | 48 hours
  blood pressure in mmhg
hemodynamic changes | 48 hours
  heart rate per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year
Access Criteria: open

REFERENCES:
- [Result] Chuan A, Lansdown A, Brick KL, Bourgeois AJG, Pencheva LB, Hue B, Goddard S, Lennon MJ, Walters A, Auyong D; Continuous Catheters in Adductor Canal versus Femoral Triangle (The CAFE study) investigators. Adductor canal versus femoral triangle anatomical locations for continuous catheter analgesia after total knee arthroplasty: a multicentre randomised controlled study. Br J Anaesth. 2019 Sep;123(3):360-367. doi: 10.1016/j.bja.2019.03.021. Epub 2019 May 2. PMID 31056239